CLINICAL TRIAL: NCT06788015
Title: The Effects of Hydrogen-Infused Water on Endurance Performance, Body Hydration Biomarkers, and Health-Related Quality of Life in Healthy Young Men and Women (HYDRO2EAU): A Randomized-Controlled Clinical Trial
Brief Title: Hydrogen-Infused Water for Endurance Performance, Body Hydration Biomarkers, and Health-Related Quality of Life
Acronym: HYDRO2EAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: THIC-1-24
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Exercise Overtraining
Keywords: endurance
MeSH Terms: conditions — Overtraining Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen-infused water (Experimental): One can of hydrogen-infused water consumed before breakfast and dinner
  Interventions: Dietary Supplement: Hydrogen-infused water
- Placebo (Placebo Comparator): One can of hydrogen-free water consumed before breakfast and dinner
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hydrogen-infused water — Water containing molecular hydrogen
  Arms: Hydrogen-infused water
Dietary Supplement: Placebo — Water containing no molecular hydrogen
  Arms: Placebo

SUMMARY:
The study investigates the impact of 4-week hydrogen-infused water consumption on various health and performance outcomes. Conducted with healthy young adults, the trial assesses endurance performance, hydration biomarkers, and health-related quality of life. Participants are randomized into intervention and control groups, with outcomes measured over a specified period. The findings aim to elucidate whether hydrogen-infused water water provides significant benefits for physical performance, hydration status, and overall well-being compared to standard hydration methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18.0 - 29.9 years
* Body mass index 18.5 - 24.9 kg/m2
* Collegiate athletes with training experience >3 years
* Weekly exercise > 5 hours
* Given written informed consent

Exclusion Criteria:

* Major chronic diseases or acute disorders
* History of dietary supplement usage in the 4 weeks preceding the study initiation
* Unwillingness to return for a follow-up
* Participation in other clinical trials

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Time to exhaustion | Change from baseline time to exhaustion at 4 weeks
  Running time to exhaustion at treadmill

SECONDARY OUTCOMES:
Total body water | Change from baseline total body water at 4 weeks
  Level of total body water

OTHER OUTCOMES:
36-Item Short Form Health Survey | Change from baseline 36-Item Short Form Health Survey total score at 4 weeks
  Short Form Health Survey total score, minimum and maximum possible score of between 0 and 100, with higher scores mean better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- FSPE Applied BIoenergetics Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in hydrogen research in biomedicine. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Ostojic SM. Hydrogen Gas as an Exotic Performance-Enhancing Agent: Challenges and Opportunities. Curr Pharm Des. 2021;27(5):723-730. doi: 10.2174/1381612826666200922155242. PMID 32962610